CLINICAL TRIAL: NCT06456970
Title: Frequency of Metabolic Dysfunction Associated Fatty Liver Disease in Patients With Acute Coronary Syndromes
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Taiseer Mohamed Kamal El Deen Hasanin Mohamed, Assistant Lecturer, Assiut University
Other Study IDs: MAFLD and ACS
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: fibroscan — Fibroscan examination with controlled attenuation parameter"CAP" (Echosens FibroScan ® Compact 530) for evaluation of steatosis and its degree (by CAP score) and fibrosis stage by liver stiffness measurement(LSM)

SUMMARY:
Aim of the research is to assess frequency of MAFLD among patients with acute coronary syndromes (ACS).

DETAILED DESCRIPTION:
Hepatic manifestation of metabolic syndrome (MS) is known as Metabolic Dysfunction Associated Fatty Liver Disease (MAFLD). MAFLD could be complicated by serious events as steatohepatitis, cirrhosis and malignant liver. The characteristics histological findings in those patients are macrovesicular steatosis. The prevalence of MAFLD has doubled over the last 20 years.

Globally, based on many reported studies, it's well-known that in 25-28% of deaths in patients with Metabolic Dysfunction Associated Fatty Liver Disease (MAFLD) , coronary artery disease (CAD) is accused to be the leading cause.

Patients with MAFLD are known to have more complex coronary artery disease in angiography. But the effect on clinical outcome and mortality is not known. Furthermore, the impact of MAFLD on acute coronary syndrome (ACS) is not clear. Moreover, in patients with metabolic syndrome the presence of MAFLD would be associated with severe form of CAD as noticed by angiography where there was increased in number of affected vessels and multivariate regression analysis found that MAFLD as the only independent factor affecting coronary score.

The SYNTAX score was prospectively developed for the SYNTAX trial to grade the anatomical complexity of coronary lesions in patients with lt main coronary arterty (LM) or three-vessel disease . It was found to be an independent predictor of long-term major adverse cardiac and cerebrovascular events (MACCE) and of death.

While the available data clearly support a role of MAFLD in initiating and progression of CAD in non-diabetic patients is still to be searched. MAFLD might play a part in the pathogenesis of CAD through the overexpression and systemic release of several inﬂammatory, hemostatic and oxidative-stress mediators or via contributing to whole-body insulin resistance and atherogenic dyslipidemia.

Based on the lack of studies that discussed the effect of MAFLD on patients with ACS ,we designed this study trying to asses the effect of MAFLD on the severity of ACS.

ELIGIBILITY:
Inclusion Criteria:

Any Patient above the age of 18 years old presented with acute coronary syndromes {myocardial infarction (MI), non-ST elevation myocardial infarction (NSTEMI), unstable angina} underwent coronary angiography within admission.

Exclusion Criteria:

1. Patients refused to participate.
2. Patients with history of alcohol or drug abuse.
3. Patients have hepatitis C or hepatitis B infection.
4. Patients have primary or secondary hepatic malignancies
5. Pregnant women.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any Patient above the age of 18 years presented with acute coronary syndromes {myocardial infarction (MI), non-ST elevation myocardial infarction (NSTEMI), unstable angina} underwent coronary angiography within admission.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Assess frequency of MAFLD among patients with acute coronary syndromes (ACS). | baseline
  patients with acute coronary syndrome will be evaluated if they have MAFLD and then we will know frequency of MAFLD among patients with acute coronary syndromes (ACS)

CONTACTS AND LOCATIONS:
Overall Officials: Taiseer Mohamed Kamal El Deen, resident, Principal Investigator — Assiut University; Waleed Attia Hassan, A.professor, Study Director — Assiut University; Sahar Mohammed Hassany, professor, Study Director — Assiut University; Mohamed Osman Abdelhameed, Lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Katsiki N, Perez-Martinez P, Anagnostis P, Mikhailidis DP, Karagiannis A. Is Nonalcoholic Fatty Liver Disease Indeed the Hepatic Manifestation of Metabolic Syndrome? Curr Vasc Pharmacol. 2018;16(3):219-227. doi: 10.2174/1570161115666170621075619. PMID 28669328
- [Background] Malnick S, Maor Y. The Interplay between Alcoholic Liver Disease, Obesity, and the Metabolic Syndrome. Visc Med. 2020 Jun;36(3):198-205. doi: 10.1159/000507233. Epub 2020 Apr 23. PMID 32775350
- [Background] Eddy DM, Schlessinger L, Heikes K. The metabolic syndrome and cardiovascular risk: implications for clinical practice. Int J Obes (Lond). 2008 May;32 Suppl 2:S5-10. doi: 10.1038/ijo.2008.28. PMID 18469838
- [Background] Huang Z, Wang X, Ding X, Cai Z, Li W, Chen Z, Fang W, Cai Z, Lan Y, Chen G, Wu W, Chen Z, Wu S, Chen Y. Association of Age of Metabolic Syndrome Onset With Cardiovascular Diseases: The Kailuan Study. Front Endocrinol (Lausanne). 2022 Mar 17;13:857985. doi: 10.3389/fendo.2022.857985. eCollection 2022. PMID 35370968
- [Background] Ren Z, Simons PIHG, Wesselius A, Stehouwer CDA, Brouwers MCGJ. Relationship between NAFLD and coronary artery disease: A Mendelian randomization study. Hepatology. 2023 Jan 1;77(1):230-238. doi: 10.1002/hep.32534. Epub 2022 May 18. PMID 35441719
- [Background] Sianos G, Morel MA, Kappetein AP, Morice MC, Colombo A, Dawkins K, van den Brand M, Van Dyck N, Russell ME, Mohr FW, Serruys PW. The SYNTAX Score: an angiographic tool grading the complexity of coronary artery disease. EuroIntervention. 2005 Aug;1(2):219-27. No abstract available. PMID 19758907
- [Background] Cavalcante R, Sotomi Y, Mancone M, Whan Lee C, Ahn JM, Onuma Y, Lemos PA, van Geuns RJ, Park SJ, Serruys PW. Impact of the SYNTAX scores I and II in patients with diabetes and multivessel coronary disease: a pooled analysis of patient level data from the SYNTAX, PRECOMBAT, and BEST trials. Eur Heart J. 2017 Jul 1;38(25):1969-1977. doi: 10.1093/eurheartj/ehx138. PMID 28431047
- [Background] Abosheaishaa H, Hussein M, Ghallab M, Abdelhamid M, Balassiano N, Ahammed MR, Baig MA, Khan J, Elshair M, Soliman MY, Abdelwahed M, Ali A, Alzamzamy A, Nassar M. Association between non-alcoholic fatty liver disease and coronary artery disease outcomes: A systematic review and meta-analysis. Diabetes Metab Syndr. 2024 Jan;18(1):102938. doi: 10.1016/j.dsx.2023.102938. Epub 2024 Jan 3. PMID 38194827
- [Background] Baharvand-Ahmadi B, Sharifi K, Namdari M. Prevalence of non-alcoholic fatty liver disease in patients with coronary artery disease. ARYA Atheroscler. 2016 Jul;12(4):201-205. PMID 28149317
- [Background] Keys A, Fidanza F, Karvonen MJ, Kimura N, Taylor HL. Indices of relative weight and obesity. J Chronic Dis. 1972 Jul 1;25(6):329-43. doi: 10.1016/0021-9681(72)90027-6. No abstract available. PMID 4650929
- [Background] WHO Expert Consultation. Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies. Lancet. 2004 Jan 10;363(9403):157-63. doi: 10.1016/S0140-6736(03)15268-3. PMID 14726171
- [Background] Eslam M, Sarin SK, Wong VW, Fan JG, Kawaguchi T, Ahn SH, Zheng MH, Shiha G, Yilmaz Y, Gani R, Alam S, Dan YY, Kao JH, Hamid S, Cua IH, Chan WK, Payawal D, Tan SS, Tanwandee T, Adams LA, Kumar M, Omata M, George J. The Asian Pacific Association for the Study of the Liver clinical practice guidelines for the diagnosis and management of metabolic associated fatty liver disease. Hepatol Int. 2020 Dec;14(6):889-919. doi: 10.1007/s12072-020-10094-2. Epub 2020 Oct 1. PMID 33006093
- See also: Is Nonalcoholic Fatty Liver Disease Indeed the Hepatic Manifestation of Metabolic Syndrome? — https://pubmed.ncbi.nlm.nih.gov/28669328/
- See also: The Interplay between Alcoholic Liver Disease, Obesity, and the Metabolic Syndrome — https://pubmed.ncbi.nlm.nih.gov/32775350/
- See also: The metabolic syndrome and cardiovascular risk: implications for clinical practice — https://pubmed.ncbi.nlm.nih.gov/18469838/
- See also: Association of Age of Metabolic Syndrome Onset With Cardiovascular Diseases: The Kailuan Study — https://pubmed.ncbi.nlm.nih.gov/35370968/
- See also: Relationship between NAFLD and coronary artery disease: A Mendelian randomization study — https://pubmed.ncbi.nlm.nih.gov/35441719/
- See also: The SYNTAX Score: an angiographic tool grading the complexity of coronary artery disease — https://pubmed.ncbi.nlm.nih.gov/19758907/
- See also: Impact of the SYNTAX scores I and II in patients with diabetes and multivessel coronary disease: a pooled analysis of patient level data from the SYNTAX, PRECOMBAT, and BEST trials — https://pubmed.ncbi.nlm.nih.gov/28431047/
- See also: Association between non-alcoholic fatty liver disease and coronary artery disease outcomes: A systematic review and meta-analysis — https://pubmed.ncbi.nlm.nih.gov/38194827/
- See also: Prevalence of non-alcoholic fatty liver disease in patients with coronary artery disease — https://pubmed.ncbi.nlm.nih.gov/28149317/
- See also: Indices of relative weight and obesity — https://pubmed.ncbi.nlm.nih.gov/4650929/
- See also: Appropriate body-mass index for Asian populations and its implications for policy and intervention strategies — https://pubmed.ncbi.nlm.nih.gov/14726171/
- See also: The Asian Pacific Association for the Study of the Liver clinical practice guidelines for the diagnosis and management of metabolic associated fatty liver disease — https://pubmed.ncbi.nlm.nih.gov/33006093/